CLINICAL TRIAL: NCT04421365
Title: Adaptive Closed-loop Brain-computer Interface Therapeutic Intervention in Laryngeal Dystonia
Brief Title: Brain-Computer Interfaces in Laryngeal Dystonia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kristina Simonyan (Other)
Responsible Party: Sponsor-Investigator, Kristina Simonyan, Professor of Otolaryngology - Head and Neck Surgery, Massachusetts Eye and Ear Infirmary
Organization: Massachusetts Eye and Ear Infirmary (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 2019P001547
Record Dates: First submitted 2020-05-15; First posted 2020-06-09 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Laryngeal Dystonia
MeSH Terms: conditions — Dysphonia

STUDY DESIGN:
Intervention Model Description: Patients will be assigned to active neurofeedback BCI and sham neurofeedback BCI groups to assess the feasibility of the BCI system and the efficacy of neurofeedback.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Active neurofeedback BCI (Active Comparator): Patients are presented with symptomatic speech and asymptomatic whisper and, using active EEG-based neurofeedback, are trained to correct their speech by matching their brain patterns to those of whisper. This training is expected to be effective for symptom improvement.
  Interventions: Device: neurofeedback brain-computer interface (BCI)
- Sham neurofeedback BCI (Sham Comparator): Patients are presented with symptomatic speech and asymptomatic whisper and, using sham EEG-based neurofeedback, are trained to correct their speech by matching their brain patterns to those of whisper. This training is expected not to be effective for symptom improvement.
  Interventions: Device: neurofeedback brain-computer interface (BCI)

INTERVENTIONS:
Device: neurofeedback brain-computer interface (BCI) — The integrated components of BCI system include the high-density EEG, 3D-VR, and a built-in ML platform as a real-time neural signal decoder and neurofeedback controller.

SUMMARY:
The researchers will develop and evaluate the use of adaptive closed-loop brain-computer interface therapeutic intervention in laryngeal dystonia.

DETAILED DESCRIPTION:
Dystonia is a neurological disorder, which causes involuntary, sustained muscle contractions, resulting in uncontrollable twisting, repetitive movements, and abnormal postures. Selective impairment of motor control of highly skilled and goal-oriented behaviors is the defining feature of task-specific focal dystonias. Among these, laryngeal dystonia (LD) is characterized by involuntary spasms in laryngeal muscles, which selectively occur during speaking but not whispering, crying, or laughing. As speech communication is a vital part of our daily existence, LD symptoms have a deeply pervasive effect on the quality of life of the affected individual, often extending beyond speech motor deficits and causing significant occupational disability, psychiatric comorbidities, long-lasting stress, and social isolation.

Despite the chronic, debilitating impact of LD, its clinical management remains stagnant. The overall objective of this study is to conduct a randomized, sham-controlled, parallel design, phase 1 clinical trial to assess the feasibility and efficacy of a neurofeedback brain-computer interface (BCI) paradigm in LD patients that acts upon and modulates the disorder pathophysiology. The rationale for the proposed studies is that delineation of task-specific neural alterations for their feasible utilization as a pathophysiological target of therapeutic intervention will establish a robust scientific foundation for the development of novel strategies for LD treatment, inform the conduct of the next phase of the clinical trial, and directly contribute to closing the existing critical gap in the clinical management of this disorder.

ELIGIBILITY:
Inclusion criteria:

1. Patients will have clinically documented isolated adductor laryngeal dystonia (ADLD) without any other forms of dystonia or tremor. ADLD causes involuntary spasms during vocal fold adduction, leading to voice breaks predominantly on vowels and strained, strangles quality of voice, predominantly affecting voice production during the speaking. Only patients with the ADLD form of disorder will be recruited to minimize the impact of heterogeneity of voice symptomatology on the outcome of these phase 1 studies;
2. Healthy controls will be healthy individuals with a negative history of any neurological, psychiatric, or laryngeal problems;
3. Age from 18 to 80 years;
4. Native English speakers. Non-English-speaking subjects will not be recruited because brain activation and neural network organization are different between native and non-native English speakers;
5. Right-handedness (based on Edinburgh Handedness Inventory). Left-handed subjects will not be recruited because brain activation and neural network organization are different between right and left-handed individuals;
6. Normal cognitive status (based on Montreal Cognitive Assessment).

Exclusion criteria:

1. Subjects who are incapable of giving informed consent will be excluded from the study;
2. Pregnant or breastfeeding women until the time they are no longer pregnant or breastfeeding will be excluded from the study. All women of childbearing potential will undergo a urine pregnancy test, which must be negative for study participation;
3. Subjects with a past or present medical history of (a) neurological problems, such as stroke, movement disorders (except for ADLD in the patient group), brain tumors, ataxias, myopathies, myasthenia gravis, demyelinating diseases; (b) psychiatric problems, such as schizophrenia, bipolar depression, obsessive-compulsive disorder; (c) laryn¬geal problems, such as vocal fold paralysis, paresis, carcinoma;
4. Subjects with impaired hearing, vision, and speaking abilities (except for ADLD), as these would most typically have a neurological origin;
5. Patients who have dystonia symptoms at rest in order to avoid the potential confound of dystonic spasms occurring during the asymptomatic task production;
6. Patients who are not symptomatic due to the treatment with botulinum toxin injections into the affected muscles. The duration of positive effects of botulinum toxin varies from patient to patient but lasts on average for 3-4 months. All patients will be evaluated to ensure that they are fully symptomatic and are at least three months post-injection prior to study participation;
7. To avoid the possibility of confounding effects of drugs acting upon the central nervous system, all subjects will be questioned about any prescribed or over-the-counter medications as part of their initial screening. Those who are on medication(s) affecting the central nervous system will be excluded;
8. Subjects with implanted deep brain stimulators will be excluded from the study;
9. Subjects will be asked whether they have undergone any head and neck surgeries, particularly any brain surgery and laryngeal surgeries, such as thyroplasty, laryngeal denervation, and selective laryngeal adductor denervation-reinnervation. Because both brain and laryngeal surgery may potentially lead to the brain structure and function re-organization, all subjects with a history of brain and/or laryngeal surgery will be excluded from the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-04-18 (Actual); Primary Completion 2027-08-31 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Changes in voice symptoms | At the end of day 5 of the intervention
  Change in the number of dystonic voice breaks as the result of active neurofeedback BCI intervention assessed using perceptual voice analysis

CONTACTS AND LOCATIONS:
Overall Officials: Kristina Simonyan, MD, PhD, Principal Investigator — Massachusetts Eye and Ear
Locations (1):
- Massachusetts Eye and Ear Infirmary, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No